CLINICAL TRIAL: NCT04958096
Title: Adjunct Cortical Stimulation With Deep Brain Stimulation (DBS) to Treat Obsessive Compulsive Disorder (OCD)
Brief Title: Cortical Stimulation to Treat Obsessive Compulsive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Moses Lee, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Andrew Moses Lee, MD, PhD, Assistant Professor, Psychiatry, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-33743
Record Dates: First submitted 2021-06-27; First posted 2021-07-12 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; Obsessive Compulsive Disorder; Obsessive thoughts; Compulsions
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Compulsive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Prefrontal Cortex (PFC) (Experimental): The Prefrontal Cortex (PFC) treatment group will be have an implant bilaterally at the HDE-approved ALIC site and the PFC.
  Interventions: Device: Standard Therapeutic Deep Brain Stimulation; Device: Cortical Stimulation for PFC
- Anterior Cingulate Cortex (ACC) (Experimental): The Anterior Cingulate Cortex (ACC) treatment group will be have an implant bilaterally at the HDE-approved ALIC site and the ACC.
  Interventions: Device: Standard Therapeutic Deep Brain Stimulation; Device: Cortical Stimulation for ACC

INTERVENTIONS:
Device: Standard Therapeutic Deep Brain Stimulation — DBS to the standard subcortical targets (anterior limb of the internal capsule- ALIC) will be used to treat OCD
Device: Cortical Stimulation for PFC — Patients enrolled in this study will have a second pair of leads placed in the prefrontal cortex (PFC) bilaterally as well the surrounding white matter tracts and stimulation will be delivered through these leads to improve OCD symptoms
  Other Names: PFC Stimulation
  Arms: Prefrontal Cortex (PFC)
Device: Cortical Stimulation for ACC — Patients enrolled in this study will have a second pair of leads placed in the anterior cingulate cortex (ACC) bilaterally as well the surrounding white matter tracts and stimulation will be delivered through these leads to improve OCD symptoms
  Other Names: OCD Cortical Stimulation
  Arms: Anterior Cingulate Cortex (ACC)

SUMMARY:
The purpose of this study is to identify abnormal brain signals associated with Obsessive Compulsive Disorder (OCD) and psychiatric symptoms and to investigate novel therapeutic stimulation sites. While treating OCD with standard deep brain stimulation (DBS) therapy, the investigators will also monitor the activity of the anterior cingulate and prefrontal cortex, a region known be involved with OCD, decision making, and emotion regulation, and the investigators will identify abnormal activity corresponding to the severity of a patient's OCD. The investigators will also investigate whether it is possible for stimulation delivered to these parts of the brain can improve OCD symptoms. These investigations have the potential to aid in the development of improved forms of DBS that can better target abnormal OCD brain signatures in the future.

The investigators will implant a cortical electrode in addition to the ALIC DBS electrode and connect these to an implantable pulse generator that care store field potential data (Medtronic Percept). The decision whether the lead is placed in the prefrontal or cingulate cortex bilaterally will be based upon considerations of the surgical risks for a particular patient based upon their anatomy and the required surgical approach.

At multiple time points post-implantation up to 2 years, in our clinic or patient's homes, cortical and subcortical signals will be recorded. Data will be collected while patient are resting or engaged in symptom provocation tasks, emotional/cognitive tasks while cortical stimulation is on and off. In addition to brain signal recordings, symptoms will be assessed using validated questionnaires and tasks to allow identification of neurophysiological correlates of OCD symptoms.

DETAILED DESCRIPTION:
The investigators propose to perform electrophysiological investigations into the corticostriatal circuits mediating severe, refractory obsessive compulsive disorder (OCD) through chronic intracranial recordings and stimulation. This new study will utilize the Medtronic Percept, which is currently is approved for treating OCD under the Humanitarian Device Exemption (HDE).

In addition to their standard therapeutic DBS electrode(s) in the standard subcortical targets (anterior limb of the internal capsule- ALIC), patients enrolled in this study will have a second pair of leads placed in either the prefrontal cortex (PFC) or anterior cingulate cortex (ACC) bilaterally as well the surrounding white matter tracts for a total of 4 DBS leads.

After electrode implantations, patient will undergo 2 phases:

In phase 1 (day 1 - 12 months), the aim will be to identify a biomarker of OCD-related symptoms. Patient will undergo long-term monitoring of their OCD and related psychiatric symptoms along with recordings of cortical and subcortical local field potentials (LFPs). This phase will be conducted in both the outpatient office setting and patient's home environment.

In phase 2 (13 months - 2 years), the investigators will introduce cortical stimulation at either the PFC or ACC/cingulum in addition to stimulation at the ALIC. The investigators will continue to obtain brain recordings and ratings during this period of time to identify the impact of cortical stimulation on these signals.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent for the study
* Age 22-75
* Clinical diagnosis of OCD
* Documented duration of OCD of at least 5 years
* OCD rated as severe or extreme illness (YBOCs ≥ 28)
* Has failed to improve following treatment with at least two selective serotonin reuptake inhibitors (SSRIs), clomipramine, and augmentation with antipsychotics
* Has not responded to adequate trials of cognitive behavior therapy (exposure and response prevention)
* Has not responded adequately to TMS treatment for OCD if it is reasonably available to the patient

Exclusion Criteria:

* Has hoarding as a primary subclassification of OCD according to DSM-4
* Has another severe psychiatric disorder (personality disorder, psychotic/bipolar disorder, etc) or substance abuse issues
* Is pregnant
* Has an abnormal MRI assessed by the team or has a neurological condition requiring an MRI in the future
* Has a cognitive disorder or dementia
* Is at imminent risk for suicide based upon Suicide Severity Rating Scale (SSRS) or has ever attempted suicide
* Inability to comply with study follow-up visits
* Major comorbidity increasing the risk of surgery (prior stroke, severe hypertension, severe diabetes, or need for chronic anticoagulation other than aspirin)
* Allergies or known hypersensitivity to materials in the Activa systems (i.e. titanium, polyurethane, silicone, polyethermide, stainless steel).
* Previous cranial ablative or deep brain stimulation surgery.
* Patients may be excluded from enrollment due to a condition that, in the judgement of the PI, significantly increases risk or reduces significantly the likelihood of benefit from DBS.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Yale-Brown Obsessive Compulsive Scale (Y-BOCS) from 12 months to 24 months | 12-24 months
  The Y-BOCS is an OCD symptom scale used for identifying current OCD symptom severity. The score ranges from 0-40, with higher scores indicating more severe OCD symptoms. The change in Y-BOCS score from 12 months to 24 months will be reported.

SECONDARY OUTCOMES:
Change in Montgomery Asberg Depression Rating Scale (MADRS) score from 12 months to 24 months | 12-24 months
  Effect size of cortical stim + ALIC DBS compared to ALIC DBS (mean difference in Montgomery Asberg Depression Rating Scale (MADRS) score at 12 months and 24 months. Higher MADRS score indicates more severe depression; the overall score ranges from 0 to 60.

OTHER OUTCOMES:
Biomarker identification in Stage 1 | 1-12 months
  The number of patients in whom we can identify a neural biomarker that accounts for a significant amount of variance in OCD symptom severity

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Lee, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Nancy Friend Pritzker Psychiatry Building, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Denys D. Pharmacotherapy of obsessive-compulsive disorder and obsessive-compulsive spectrum disorders. Psychiatr Clin North Am. 2006 Jun;29(2):553-84, xi. doi: 10.1016/j.psc.2006.02.013. PMID 16650723
- [Background] Denys D, Graat I, Mocking R, de Koning P, Vulink N, Figee M, Ooms P, Mantione M, van den Munckhof P, Schuurman R. Efficacy of Deep Brain Stimulation of the Ventral Anterior Limb of the Internal Capsule for Refractory Obsessive-Compulsive Disorder: A Clinical Cohort of 70 Patients. Am J Psychiatry. 2020 Mar 1;177(3):265-271. doi: 10.1176/appi.ajp.2019.19060656. Epub 2020 Jan 7. PMID 31906709
- [Background] Swann NC, de Hemptinne C, Thompson MC, Miocinovic S, Miller AM, Gilron R, Ostrem JL, Chizeck HJ, Starr PA. Adaptive deep brain stimulation for Parkinson's disease using motor cortex sensing. J Neural Eng. 2018 Aug;15(4):046006. doi: 10.1088/1741-2552/aabc9b. Epub 2018 May 9. PMID 29741160
- [Background] Starr PA. Totally Implantable Bidirectional Neural Prostheses: A Flexible Platform for Innovation in Neuromodulation. Front Neurosci. 2018 Sep 7;12:619. doi: 10.3389/fnins.2018.00619. eCollection 2018. PMID 30245616
- [Background] Dougherty DD, Brennan BP, Stewart SE, Wilhelm S, Widge AS, Rauch SL. Neuroscientifically Informed Formulation and Treatment Planning for Patients With Obsessive-Compulsive Disorder: A Review. JAMA Psychiatry. 2018 Oct 1;75(10):1081-1087. doi: 10.1001/jamapsychiatry.2018.0930. PMID 30140845
- [Background] Milad MR, Rauch SL. Obsessive-compulsive disorder: beyond segregated cortico-striatal pathways. Trends Cogn Sci. 2012 Jan;16(1):43-51. doi: 10.1016/j.tics.2011.11.003. Epub 2011 Dec 2. PMID 22138231
- [Background] Anticevic A, Hu S, Zhang S, Savic A, Billingslea E, Wasylink S, Repovs G, Cole MW, Bednarski S, Krystal JH, Bloch MH, Li CS, Pittenger C. Global resting-state functional magnetic resonance imaging analysis identifies frontal cortex, striatal, and cerebellar dysconnectivity in obsessive-compulsive disorder. Biol Psychiatry. 2014 Apr 15;75(8):595-605. doi: 10.1016/j.biopsych.2013.10.021. Epub 2013 Nov 4. PMID 24314349
- [Background] Saxena S, Brody AL, Maidment KM, Dunkin JJ, Colgan M, Alborzian S, Phelps ME, Baxter LR Jr. Localized orbitofrontal and subcortical metabolic changes and predictors of response to paroxetine treatment in obsessive-compulsive disorder. Neuropsychopharmacology. 1999 Dec;21(6):683-93. doi: 10.1016/S0893-133X(99)00082-2. PMID 10633474
- [Background] Nabeyama M, Nakagawa A, Yoshiura T, Nakao T, Nakatani E, Togao O, Yoshizato C, Yoshioka K, Tomita M, Kanba S. Functional MRI study of brain activation alterations in patients with obsessive-compulsive disorder after symptom improvement. Psychiatry Res. 2008 Aug 30;163(3):236-47. doi: 10.1016/j.pscychresns.2007.11.001. Epub 2008 Jul 29. PMID 18667293
- [Background] Saxena S, Rauch SL. Functional neuroimaging and the neuroanatomy of obsessive-compulsive disorder. Psychiatr Clin North Am. 2000 Sep;23(3):563-86. doi: 10.1016/s0193-953x(05)70181-7. PMID 10986728
- [Background] Brown LT, Mikell CB, Youngerman BE, Zhang Y, McKhann GM 2nd, Sheth SA. Dorsal anterior cingulotomy and anterior capsulotomy for severe, refractory obsessive-compulsive disorder: a systematic review of observational studies. J Neurosurg. 2016 Jan;124(1):77-89. doi: 10.3171/2015.1.JNS14681. Epub 2015 Aug 7. PMID 26252455
- [Background] Carmi L, Tendler A, Bystritsky A, Hollander E, Blumberger DM, Daskalakis J, Ward H, Lapidus K, Goodman W, Casuto L, Feifel D, Barnea-Ygael N, Roth Y, Zangen A, Zohar J. Efficacy and Safety of Deep Transcranial Magnetic Stimulation for Obsessive-Compulsive Disorder: A Prospective Multicenter Randomized Double-Blind Placebo-Controlled Trial. Am J Psychiatry. 2019 Nov 1;176(11):931-938. doi: 10.1176/appi.ajp.2019.18101180. Epub 2019 May 21. PMID 31109199
- [Background] Nauczyciel C, Le Jeune F, Naudet F, Douabin S, Esquevin A, Verin M, Dondaine T, Robert G, Drapier D, Millet B. Repetitive transcranial magnetic stimulation over the orbitofrontal cortex for obsessive-compulsive disorder: a double-blind, crossover study. Transl Psychiatry. 2014 Sep 9;4(9):e436. doi: 10.1038/tp.2014.62. PMID 25203167
- [Background] Rao VR, Sellers KK, Wallace DL, Lee MB, Bijanzadeh M, Sani OG, Yang Y, Shanechi MM, Dawes HE, Chang EF. Direct Electrical Stimulation of Lateral Orbitofrontal Cortex Acutely Improves Mood in Individuals with Symptoms of Depression. Curr Biol. 2018 Dec 17;28(24):3893-3902.e4. doi: 10.1016/j.cub.2018.10.026. Epub 2018 Nov 29. PMID 30503621
- [Background] Sani OG, Yang Y, Lee MB, Dawes HE, Chang EF, Shanechi MM. Mood variations decoded from multi-site intracranial human brain activity. Nat Biotechnol. 2018 Nov;36(10):954-961. doi: 10.1038/nbt.4200. Epub 2018 Sep 10. PMID 30199076
- [Background] Bijanki KR, Manns JR, Inman CS, Choi KS, Harati S, Pedersen NP, Drane DL, Waters AC, Fasano RE, Mayberg HS, Willie JT. Cingulum stimulation enhances positive affect and anxiolysis to facilitate awake craniotomy. J Clin Invest. 2019 Mar 1;129(3):1152-1166. doi: 10.1172/JCI120110. Epub 2019 Feb 11. PMID 30589643
- [Background] Swann NC, de Hemptinne C, Miocinovic S, Qasim S, Ostrem JL, Galifianakis NB, Luciano MS, Wang SS, Ziman N, Taylor R, Starr PA. Chronic multisite brain recordings from a totally implantable bidirectional neural interface: experience in 5 patients with Parkinson's disease. J Neurosurg. 2018 Feb;128(2):605-616. doi: 10.3171/2016.11.JNS161162. Epub 2017 Apr 14. PMID 28409730
- [Background] Shirvalkar P, Veuthey TL, Dawes HE, Chang EF. Closed-Loop Deep Brain Stimulation for Refractory Chronic Pain. Front Comput Neurosci. 2018 Mar 26;12:18. doi: 10.3389/fncom.2018.00018. eCollection 2018. PMID 29632482
- [Background] De Ridder D, Leong SL, Manning P, Vanneste S, Glue P. Anterior Cingulate Implant for Obsessive-Compulsive Disorder. World Neurosurg. 2017 Jan;97:754.e7-754.e16. doi: 10.1016/j.wneu.2016.10.046. Epub 2016 Oct 15. PMID 27756670
- [Background] Burguiere E, Monteiro P, Feng G, Graybiel AM. Optogenetic stimulation of lateral orbitofronto-striatal pathway suppresses compulsive behaviors. Science. 2013 Jun 7;340(6137):1243-6. doi: 10.1126/science.1232380. PMID 23744950
- [Background] Pinhal CM, van den Boom BJG, Santana-Kragelund F, Fellinger L, Bech P, Hamelink R, Feng G, Willuhn I, Feenstra MGP, Denys D. Differential Effects of Deep Brain Stimulation of the Internal Capsule and the Striatum on Excessive Grooming in Sapap3 Mutant Mice. Biol Psychiatry. 2018 Dec 15;84(12):917-925. doi: 10.1016/j.biopsych.2018.05.011. Epub 2018 May 23. PMID 29954580
- [Background] Greenberg BD, Gabriels LA, Malone DA Jr, Rezai AR, Friehs GM, Okun MS, Shapira NA, Foote KD, Cosyns PR, Kubu CS, Malloy PF, Salloway SP, Giftakis JE, Rise MT, Machado AG, Baker KB, Stypulkowski PH, Goodman WK, Rasmussen SA, Nuttin BJ. Deep brain stimulation of the ventral internal capsule/ventral striatum for obsessive-compulsive disorder: worldwide experience. Mol Psychiatry. 2010 Jan;15(1):64-79. doi: 10.1038/mp.2008.55. Epub 2008 May 20. PMID 18490925
- [Background] Swann NC, de Hemptinne C, Miocinovic S, Qasim S, Wang SS, Ziman N, Ostrem JL, San Luciano M, Galifianakis NB, Starr PA. Gamma Oscillations in the Hyperkinetic State Detected with Chronic Human Brain Recordings in Parkinson's Disease. J Neurosci. 2016 Jun 15;36(24):6445-58. doi: 10.1523/JNEUROSCI.1128-16.2016. PMID 27307233
- [Background] Brown JA, Barbaro NM. Motor cortex stimulation for central and neuropathic pain: current status. Pain. 2003 Aug;104(3):431-435. doi: 10.1016/S0304-3959(03)00209-4. No abstract available. PMID 12927615
- [Background] Brown JA, Lutsep H, Cramer SC, Weinand M. Motor cortex stimulation for enhancement of recovery after stroke: case report. Neurol Res. 2003 Dec;25(8):815-8. doi: 10.1179/016164103771953907. PMID 14669524
- [Background] Panov F, Kopell BH. Use of cortical stimulation in neuropathic pain, tinnitus, depression, and movement disorders. Neurotherapeutics. 2014 Jul;11(3):564-71. doi: 10.1007/s13311-014-0283-0. PMID 24888372
- [Background] Kimmelman J, Duckworth K, Ramsay T, Voss T, Ravina B, Emborg ME. Risk of surgical delivery to deep nuclei: a meta-analysis. Mov Disord. 2011 Jul;26(8):1415-21. doi: 10.1002/mds.23770. Epub 2011 May 14. PMID 21574186
- [Background] Panov F, Levin E, de Hemptinne C, Swann NC, Qasim S, Miocinovic S, Ostrem JL, Starr PA. Intraoperative electrocorticography for physiological research in movement disorders: principles and experience in 200 cases. J Neurosurg. 2017 Jan;126(1):122-131. doi: 10.3171/2015.11.JNS151341. Epub 2016 Feb 26. PMID 26918474